CLINICAL TRIAL: NCT01577082
Title: A 12-week, Multinational, Multicentre, Randomised, Double-blind, Double-dummy, 2-arm Parallel Group Study Comparing the Efficacy and Safety of CHF 1535 200/6µg Versus Beclomethasone Dipropionate in Adult Asthmatic Patients Not Adequately Controlled on High Dose of Inhaled Corticosteroids or on Medium Dose of Inhaled Corticosteroids Plus Long-acting β2 Agonists
Brief Title: Efficacy and Safety of CHF 1535 200/6µg in Not Adequately Controlled Asthmatic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-1005-PR-0040; 2010-020602-14 (EudraCT Number)
Record Dates: First submitted 2012-04-06; First posted 2012-04-13 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Asthma
Keywords: Adults, not adequately controlled, pre-dose morning PEF
MeSH Terms: conditions — Asthma | interventions — alpha-ketoisovalerate dehydrogenase phosphatase; Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHF 1535 200/6µg (Experimental)
  Interventions: Drug: CHF1535 200/6 µg
- BDP 100µg (Active Comparator)
  Interventions: Drug: BDP 100 µg

INTERVENTIONS:
Drug: CHF1535 200/6 µg — CHF 1535 (BDP/FF) 800/24 µg daily during 12 weeks
  Arms: CHF 1535 200/6µg
Drug: BDP 100 µg — Beclomethasone Dipropionate 800µg daily during 12 weeks
  Other Names: Qvar
  Arms: BDP 100µg

SUMMARY:
The purpose of this study is to show the superiority of CHF 1535 (BDP/FF) pMDI over BDP HFA pMDI in terms of lung function considering change from baseline to the entire treatment period in average pre-dose morning PEF in adult asthmatic patients not adequately controlled on high doses of ICS or on medium dose of ICS+LABA.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female patients aged > 18 years.
* Patients with persistent asthma not optimally controlled (GINA 2010) on high doses of ICS or medium dose of ICS+LABA at a stable dose for at least 4 weeks prior to screening.
* Patients with FEV1 >= 40% and < 80% of predicted for the patient normal value and at least 0.9 L.
* Patients with a documented positive response to the reversibility test, defined as ΔFEV1 >= 12% and >= 200 mL over baseline, within 30 minutes after administration of 400 μg of salbutamol pMDI.
* At screening and at the end of the run-in period, patients with not adequately controlled asthma according to GINA 2010 and with score at the Asthma Control Questionnaire (ACQ)> 0.75

Main Exclusion Criteria:

* History of near fatal asthma or of a past hospitalisation for asthma in Intensive Care Unit or of frequent exacerbations (3 or more asthma exacerbations/ year).
* Hospitalisation, Emergency Room admission or use of systemic steroids (more than 3 days) for asthma exacerbation in the 4 weeks prior to screening visit and during the run-in period.
* Symptomatic infection of the lower airways in the 4 weeks before the screening visit.
* Current or ex-smokers with total cumulative exposure equal or more than 5 pack-years and /or having stopped smoking one year or less prior to screening visit.
* Patients with a clinically significant abnormality at 12-lead ECG or presenting a QTcB interval value in ECG > 450 msec in males or > 470 msec in females).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Pre-dose morning PEF | 12 weeks
  Change from baseline to the entire treatment period in average pre-dose morning PEF

SECONDARY OUTCOMES:
Pre-dose morning FEV1 | 2 weeks
  Change from baseline in pre-dose morning FEV1 every two weeks over a 12-week period
Asthma symptoms | 12 weeks
  Asthma symptoms collected day and night-time
Adverse Events | 14 weeks
  Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Pierluigi Paggiaro, MD, PhD, Principal Investigator — Cardio-Thoracic and Vascular Dept, University of Pisa
Locations (1):
- Cardio-Thoracic and Vascular Dept, University of Pisa, Pisa, Italy

REFERENCES:
- [Result] Paggiaro P, Corradi M, Latorre M, Raptis H, Muraro A, Gessner C, Siergiejko Z, Scuri M, Petruzzelli S. High strength extrafine pMDI beclometasone/formoterol (200/6 mug) is effective in asthma patients not adequately controlled on medium-high dose of inhaled corticosteroids. BMC Pulm Med. 2016 Dec 9;16(1):180. doi: 10.1186/s12890-016-0335-9. PMID 27938358
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2010-020602-14
- See also: CSR Synopsis available in the CHIESI Clinical Study Register — https://www.chiesi.com/clinic/CSR_Synopsis_CCD-1005-PR-0040.pdf